CLINICAL TRIAL: NCT05295641
Title: American Registry of Ambulatory or Acutely Decompensated Heart Failure
Acronym: AMERICCAASS
Status: Completed | Type: Observational
Sponsor: Fundacion Clinica Valle del Lili (Other)
Collaborators: Sociedad Interamericana de Cardiología (SIAC) (Unknown); Consejo Interamericano de Falla Cardíaca e Hipertensión Pulmonar (CIFACAH) (Unknown)
Responsible Party: Principal Investigator, Juan Esteban Gomez, Chief of the Cardiology Department, Fundacion Clinica Valle del Lili
Other Study IDs: FVL-1310
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Acute Heart Failure (AHF); Chronic Heart Failure
Keywords: Decompensated; Outpatient; Treatment; Hospitalization; Mortality; Heart Failure; Americas; Registry; Inpatient
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to better characterize and understand the population of patients with ambulatory or acutely decompensated heart failure in the American continent, getting to know their sociodemographic, clinical and paraclinical characteristics

DETAILED DESCRIPTION:
An observational, prospective and multicenter study in which ambulatory patients with a confirmed diagnosis of heart failure and those admitted to the hospitalization service due to an episode of acutely decompensated heart failure will be invited to participate in order to better characterize this population

Participants who meet the eligibility criteria will be evaluated at the moment of recruitment. Follow-ups will be performed at 1, 6 and 12 months after the initial registry for hospitalized patients. For ambulatory patients follow-up will only be performed at 12 months. These initial evaluations and subsequents follow-ups will be carried out using a standardized form for the collection of hospital and outpatient data through an electronic platform

The purpose of this study is to know sociodemographic, clinical (clinical presentation, hemodynamic profiles, in-hospital and outpatient management, re-hospitalization rate, proportion of mortality, cumulative survival and heart failure readmission-free survival) and paraclinical characteristics of this population

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older and one of the following:
* Hospitalized patient with admission diagnosis of acutely decompensated heart failure or
* Outpatient with confirmed diagnosis (main or complementary) of heart failure

Exclusion Criteria:

* Hospitalized patient with principal diagnosis of another cardiovascular / non-cardiovascular pathology and who develops an acute decompensation of heart failure during hospitalization.
* Patient on heart transplant waiting list
* Patient who has implanted or is in process of implanting a long-term ventricular assist device (eg, Heart Mate II, Heart Mate III) as a target therapy or bridge therapy to other therapies
* Patient in whom palliative management has been previously defined for his/her cardiac condition (i.e. Heart failure) or for another associated medical condition (cancer, chronic obstructive pulmonary disease (COPD), etc.)
* Patient who is discharged or referred to another institution within 48 hours of hospital stay
* Inability to comply with programmed follow-ups (telephone or in person) due to social, personal or other conditions considered by the principal investigator
* Life expectancy less than 6 months given a condition other than heart failure (Cancer, COPD, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with either ambulatory diagnosis or an acute decompensation
Sampling Method: Non-Probability Sample
Enrollment: 6732 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Characteristics of population with diagnosis of heart failure in America | Baseline
  Sociodemographic characteristics of patients with heart failure
Characteristics of population with diagnosis of heart failure in America | Baseline, at Month 1, Month 6 and Month 12
  Clinical and paraclinical characteristics of patients with heart failure

SECONDARY OUTCOMES:
Outpatient management of heart failure | Baseline and at Month 12
  Describe the ambulatory/outpatient management of patients with heart failure
Relation between outpatient treatment of heart failure with proportion of hospitalization and mortality | Baseline and at Month 12
  Relate outpatient pharmacological treatment with the proportion of hospitalization and mortality
Clinical and hemodynamic presentation of acutely decompensated heart failure | Baseline
  Describe the clinical and hemodynamic presentation of patients with acute decompensated heart failure
In-hospital management of acutely decompensated heart failure | Baseline
  Describe the in-hospital management of patients with acutely decompensated heart failure
Proportion of in-hospital mortality related with acute decompensation of heart failure | Baseline
  Determine the proportion of in-hospital mortality related with acute decompensation of heart failure
Proportion of rehospitalization at 1, 6, 12 months after hospital discharge | Month 1, Month 6 and Month 12
  Determine the proportion of rehospitalization at 1, 6 and 12 months after hospital discharge
Proportion of mortality at 1, 6, 12 months after hospital discharge | Month 1, Month 6 and Month 12
  Determine the proportion of mortality at 1, 6 and 12 months after hospital discharge
Relation between hemodynamic profile of decompensation with proportion of mortality at 1, 6, 12 months after hospital discharge | Baseline, Month 1, Month 6 and Month 12
  Relate the hemodynamic profile of decompensation with the proportion of in-hospital and ambulatory mortality at 1, 6 and 12 months after hospital discharge.
Relation between in-hospital pharmacological treatment with mortality at 1, 6, 12 months after hospital discharge | Month 1, Month 6 and Month 12
  Relate hospital pharmacological treatment with inpatient and outpatient mortality at 1, 6 and 12 months after hospital discharge.
Relation between in-hospital pharmacological treatment with proportion of readmissions at 1, 6, 12 months after hospital discharge | Month 1, Month 6 and Month 12
  Relate hospital pharmacological treatment with the proportion of readmissions at 1, 6 and 12 months after hospital discharge.
Relation between outpatient pharmacological treatment with proportion of hospitalization and mortality at 1, 6, 12 months after hospital discharge | Month 1, Month 6 and Month 12
  Relate outpatient pharmacological treatment with the proportion of hospitalization and mortality at 1, 6 and 12 months after hospital discharge.
Differences among heart failure treatment considering sociodemographic characteristics | Baseline
  Describe the differences among inpatient and outpatient treatment taking into account different demographic characteristics such as: gender, age, comorbidities, among others
Differences among proportion of rehospitalization and heart failure mortality considering sociodemographic characteristics | Baseline
  Describe the differences in the proportion of rehospitalization, hospital and outpatient mortality, taking into account different demographic characteristics: gender, age, comorbidities, among others
Differences among proportion of rehospitalization and heart failure mortality considering implementation of optimal medical treatment | Baseline, Month 1, Month 6 and Month 12
  Describe the differences in the proportion of rehospitalization, hospital and outpatient mortality, taking into account the implementation of optimal or recommended medical treatment in national and international guidelines
Differences among hospitalization and heart failure mortality considering the use of cardiac devices | Baseline, Month 1, Month 6 and Month 12
  Describe the differences between hospitalization and outpatient mortality taking into account the use of cardiac devices (cardiac resynchronization and/or implantable cardiac defibrillator) recommended in international guidelines
Cumulative heart failure survival and readmission-free survival | Baseline, Month 1, Month 6 and Month 12
  Evaluate cumulative survival and heart failure readmission-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Juan E Gomez-Mesa, MD, Principal Investigator — Fundacion Clinica Valle del Lili; Mario Speranza, MD, Principal Investigator — Hospital Clínica Bíblica; Eduardo R. Perna, MD, Principal Investigator — Instituto De Cardiología J. F. Cabral; Víctor A. Rossel, MD, Principal Investigator — Instituto Nacional del Tórax; Daniel Quesada, MD, Principal Investigator — Hospital San Vicente de Paul; Mark H. Drazner, MD, Principal Investigator — University of Texas Southwestern Medical Center; Alexander Romero, MD, Principal Investigator — Hospital Santo Tomas; Walter Alarco, MD, Principal Investigator — Instituto Nacional Cardiovascular INCOR; Sebastian Seni-Molina, MD, Principal Investigator — Fundación Valle del Lili - Registry Coordinator
Locations (119):
- United States (2):
  - North Shore University Hospital, Nothwell Health, Manhasset, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Argentina (16):
  - Sanatorio Modelo Quilmes, Quilmes, Buenos Aires
  - Sanatorio de la Trinidad Quilmes y Centro Gallego, Quilmes, Buenos Aires
  - Hospital Italiano de Córdoba, Córdoba, Córdoba Province
  - Clinica Vrsalovic / Clinica del Angelo, Formosa, Formosa Province
  - Establecimiento Asistencial Gobernador Centeno, Santa Rosa, La Pampa Province
  - Hospital San Bernardo, Salta, Salta Province
  - Clínica El Castaño - CIMAC, San Juan, San Juan Province
  - Clínica CERHU / Hospital Central Ramón Carrillo, San Luis, San Luis Province
  - Instituto Cardiovascular del Rosario, Rosario, Santa Fe Province
  - Sanatorio Santa Clara Talar, Buenos Aires
  - Hospital General de Agudos Carlos G. Durand, Buenos Aires
  - Instituto de Cardiología Juana Francisca Cabral Bolívar, Corrientes
  - Hospital Privado Universitario de Córdoba, Córdoba
  - Instituto Modelo de Cardiología Privado SRL, Córdoba
  - Hospital Descentralizado Dr. Guillermo Rawson, San Juan
  - Hospital Público Dr. Marcial V. Quiroga, San Juan
- Bolivia (2):
  - Hospital Universitario Japonés, Santa Cruz de la Sierra, Santa Cruz Department
  - Caja Petrolera de Salud, Santa Cruz de la Sierra
- Instituto Nacional del Tórax, Santiago, Chile
- Colombia (17):
  - Clinica Cardio VID, Medellín, Antioquia
  - Sociedad Clínica Iberoamericana, Barranquilla, Atlántico
  - Instituto Todo Por El Corazón, Manizales, Caldas Department
  - Clínica del Occidente, Bogotá, Cundinamarca
  - Fundación Cardioinfantil, Bogotá, Cundinamarca
  - Fundación Santa Fé de Bogotá, Bogotá, Cundinamarca
  - Hospicardio, Montería, Departamento de Córdoba
  - Unimedic Ips, Pasto, Departamento de Nariño
  - Clínica Medilaser Florencia, Florencia, Departamento del Caquetá
  - Instituto Grupsalud, Santa Marta, Magdalena Department
  - Clínica los Rosales S.A. - Centro Médico para el Corazón, Pereira, Risaralda Department
  - Fundación Cardiovascular de Colombia, Floridablanca, Santander Department
  - Clinica Avidanti S.A.S, Ibagué, Tolima Department
  - Fundación Valle del Lili, Cali, Valle del Cauca Department
  - Clínica General del Norte, Barranquilla
  - Hospital Santa Clara, Bogotá
  - Sociedad Cardiológica Colombiana S.A.S., Villavicencio
- Costa Rica (3):
  - Hospital San Vicente de Paúl, Heredia
  - Hospital Clínica Bíblica, San José
  - Hospital México, CCSS, San José
- Cuba (17):
  - Hospital Clinico Quirurgico Docente Ivan Portuondo, San Antonio de los Baños, Artemisa
  - Instituto de Cardiología y Cirugía Cardiovascular, La Habana, Departamento Occidental
  - Hospital Provincial Clinico Quirurgico Docente Leon Cuervo Rubio, Pinar del Río, Provincia de Pinar del Río
  - Hospital Provincial Clínico Quirúrgico Docente Carlos Manuel De Céspedes, Bayamo
  - Hospital Provincial Clínico Quirúrgico Docente Manuel Ascunce Domenech, Camagüey
  - Hospital Provincial Dr. Antonio Luaces Iraola, Ciego de Ávila
  - Hospital General Orlando Pantoja Tamayo, Contramaestre
  - Hospital Clínico Quirúrgico Docente Calixto García Íñiguez, La Habana
  - Hospital Clínico Quirúrgico Docente Dr. Enrique Cabrera, La Habana
  - Hospital Provincial Camilo Cienfuegos, La Habana
  - Hospital General Docente Dr. Ernesto Guevara De La Serna, Las Tunas
  - Hospital Provincial Clínico Quirúrgico Docente Cmte. Faustino Pérez, Matanzas
  - Hospital Clínico Quirúrgico Docente Héroes Del Baire, Nueva Gerona
  - Hospital Provincial Docente Marting Chang Puga, Nuevitas
  - Hospital Provincial Clínico Quirúrgico Docente Abel Santamaría, Pinar del Río
  - Cardiocentro Santiago de Cuba, Santiago de Cuba
  - Hospital Provincial Saturnino Lora, Santiago de Cuba
- Dominican Republic (4):
  - Clínica Universitaria Unión Médica del Norte, Santiago de los Caballeros, Santiago Province
  - Hospital Regional Presidente Estrella Ureña, Santiago de los Caballeros, Santiago Province
  - Centro Médico Siglo 21, San Francisco de Macorís
  - Hospital Metropolitano de Santiago Homs, Santiago de los Caballeros
- Ecuador (10):
  - Hospital Luis Vernaza, Guayaquil, Guayas
  - Hospital Clínica Kennedy, Guayaquil, Guayas
  - Centro Médico de Especialidades Ameds, Manta, Manabí
  - HOSPICOR, Manta, Manabí
  - Centro Cardiológico A.C.I, Portoviejo, Manabí
  - Hospital Metropolitano, Quito, Pichincha
  - Hospital José Carrasco Arteaga / Instituto ecuatoriano de seguridad social, Cuenca
  - Clinica Jesús De Nazareth / Hospital San Marcos, Machala
  - Hospital General EISS Portoviejo, Portoviejo
  - Centro De Diagnóstico Y Tratamiento De Enfermedades (Cdt) Cardiovasculares Cardioheredia, Samborondón
- El Salvador (3):
  - Clínica de Cardiología y Ortopedia CCO, San Salvador, San Salvador Department
  - Instituto Salvadoreño del Seguro Social, San Salvador, San Salvador Department
  - Clínica del Corazón Sinusal, San Salvador
- Guatemala (5):
  - Hospital General San Juan de Dios, Guatemala City, Departamento de Guatemala
  - Hospital Roosevelt, Guatemala City, Departamento de Guatemala
  - Clínicas HART y Hospital Regional de Occidente, Quetzaltenango, Departamento de Quetzaltenango
  - Cardiocentro Chimaltenango, Chimaltenango
  - Hospital Regional de Zacapa, Zacapa
- Honduras (2):
  - Cardio Medical Center, Tegucigalpa, Francisco Morazán Department
  - Instituto Nacional Cardiopulmonar, Tegucigalpa, Francisco Morazán Department
- Heart institute of the caribbean, Kingston, Jamaica
- Mexico (7):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes, Aguascalientes
  - Christus Muguerza Hospital Alta Especialidad, Monterrey, Nuevo León
  - Hospital Español. Sociedad de Beneficencia Española I.A.P, Mexico City
  - Instituto Nacional de Cardiología Ignacio Chávez, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran, Mexico City
  - Servicios Profesionales Del Sagrado Corazón De Jesús S.C., Mexico City
  - TecSalud, Escuela de Medicina y Ciencias de la Salud del ITESM, Monterrey
- Hospital Carlos R Huembes/Clinica Plaza España/Clinica Centro Medico Juigalpa, Managua, Nicaragua
- Hospital Santo Tomás, Panama City, Panama
- Paraguay (8):
  - Hospital Nacional de Itaugua, Itauguá, Central Department
  - Hospital Central - Instituto de Previsión Social, Asunción
  - Instituto Nacional de Cardiología "Prof. Dr. Juan A. Catonni", Asunción
  - Instituto Cardiovascular del Sanatorio Migone, Asunción
  - Sanatorio Adventista de Asunción, Asunción
  - Sanatorio Italiano, Asunción
  - Clinicor Estudios Cardiológicos, Concepción
  - Hospital de Clínicas - Facultad de ciencias médicas, San Lorenzo
- Peru (6):
  - Hospital III EsSalud Chimbote, Chimbote, Ancash
  - Luis Heysen Inchaustegui - ESSALUD, Chiclayo
  - Hospital María Auxiliadora, Lima
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Nacional Daniel Alcides Carrión, Lima
  - Instituto Cardiovascular Clinicor Norte, Lima
- Thorax Centrum Paramaribo /Academic Hospital Paramaribo, Paramaribo, Suriname
- Uruguay (2):
  - Hospital de Clínicas Doctor Manuel Quintela, Montevideo
  - Médica Uruguaya, Montevideo
- Venezuela (10):
  - Clínica Chilemex, Puerto Ordaz and San Felix, Bolívar
  - Unidad Cardiovascular Ferrer, Puerto Cabello, Carabobo
  - Centro Policlínico Valencia, Valencia, Carabobo
  - ASCARDIO, Barquisimeto, Lara
  - Instituto Autónomo Hospital Universitario de Los Andes, Mérida, Mérida
  - Centro Clinico Santa Rosa, Cumaná, Sucre
  - Cardiología Tropical Azoátegui, Anzoátegui
  - Atimed C.A, Cumaná
  - IVSS Hospital Dr. Rafael Calles Sierra, Punto Fijo
  - Unicor/Funvic, Valencia

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD, since we are not allowed to share information concerning medical history of our patients

REFERENCES:
- [Background] Adams KF Jr, Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP; ADHERE Scientific Advisory Committee and Investigators. Characteristics and outcomes of patients hospitalized for heart failure in the United States: rationale, design, and preliminary observations from the first 100,000 cases in the Acute Decompensated Heart Failure National Registry (ADHERE). Am Heart J. 2005 Feb;149(2):209-16. doi: 10.1016/j.ahj.2004.08.005. PMID 15846257
- [Background] Jonsson A, Edner M, Alehagen U, Dahlstrom U. Heart failure registry: a valuable tool for improving the management of patients with heart failure. Eur J Heart Fail. 2010 Jan;12(1):25-31. doi: 10.1093/eurjhf/hfp175. PMID 20023041
- [Background] McMurray JJ, Stewart S. Epidemiology, aetiology, and prognosis of heart failure. Heart. 2000 May;83(5):596-602. doi: 10.1136/heart.83.5.596. No abstract available. PMID 10768918
- [Background] Mosterd A, Hoes AW. Clinical epidemiology of heart failure. Heart. 2007 Sep;93(9):1137-46. doi: 10.1136/hrt.2003.025270. PMID 17699180
- [Background] Hernandez-Leiva E. [Epidemiology of acute coronary syndrome and heart failure in Latin America]. Rev Esp Cardiol. 2011 Jul;64 Suppl 2:34-43. doi: 10.1016/j.recesp.2011.01.022. Spanish. PMID 21807285
- [Background] Bocchi EA, Arias A, Verdejo H, Diez M, Gomez E, Castro P; Interamerican Society of Cardiology. The reality of heart failure in Latin America. J Am Coll Cardiol. 2013 Sep 10;62(11):949-58. doi: 10.1016/j.jacc.2013.06.013. Epub 2013 Jul 10. PMID 23850910
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P. 2016 ESC Guidelines for the Diagnosis and Treatment of Acute and Chronic Heart Failure. Rev Esp Cardiol (Engl Ed). 2016 Dec;69(12):1167. doi: 10.1016/j.rec.2016.11.005. No abstract available. English, Spanish. PMID 27894487
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Background] Brouwers FP, de Boer RA, van der Harst P, Voors AA, Gansevoort RT, Bakker SJ, Hillege HL, van Veldhuisen DJ, van Gilst WH. Incidence and epidemiology of new onset heart failure with preserved vs. reduced ejection fraction in a community-based cohort: 11-year follow-up of PREVEND. Eur Heart J. 2013 May;34(19):1424-31. doi: 10.1093/eurheartj/eht066. Epub 2013 Mar 6. PMID 23470495
- [Background] Lam CS, Donal E, Kraigher-Krainer E, Vasan RS. Epidemiology and clinical course of heart failure with preserved ejection fraction. Eur J Heart Fail. 2011 Jan;13(1):18-28. doi: 10.1093/eurjhf/hfq121. Epub 2010 Aug 3. PMID 20685685
- [Background] Levy D, Kenchaiah S, Larson MG, Benjamin EJ, Kupka MJ, Ho KK, Murabito JM, Vasan RS. Long-term trends in the incidence of and survival with heart failure. N Engl J Med. 2002 Oct 31;347(18):1397-402. doi: 10.1056/NEJMoa020265. PMID 12409541
- [Background] Roger VL, Weston SA, Redfield MM, Hellermann-Homan JP, Killian J, Yawn BP, Jacobsen SJ. Trends in heart failure incidence and survival in a community-based population. JAMA. 2004 Jul 21;292(3):344-50. doi: 10.1001/jama.292.3.344. PMID 15265849
- [Background] Barker WH, Mullooly JP, Getchell W. Changing incidence and survival for heart failure in a well-defined older population, 1970-1974 and 1990-1994. Circulation. 2006 Feb 14;113(6):799-805. doi: 10.1161/CIRCULATIONAHA.104.492033. Epub 2006 Feb 6. PMID 16461823
- [Background] Jhund PS, Macintyre K, Simpson CR, Lewsey JD, Stewart S, Redpath A, Chalmers JW, Capewell S, McMurray JJ. Long-term trends in first hospitalization for heart failure and subsequent survival between 1986 and 2003: a population study of 5.1 million people. Circulation. 2009 Feb 3;119(4):515-23. doi: 10.1161/CIRCULATIONAHA.108.812172. Epub 2009 Jan 19. PMID 19153268
- [Background] Levy D, Larson MG, Vasan RS, Kannel WB, Ho KK. The progression from hypertension to congestive heart failure. JAMA. 1996 May 22-29;275(20):1557-62. PMID 8622246
- [Background] Ho KK, Pinsky JL, Kannel WB, Levy D. The epidemiology of heart failure: the Framingham Study. J Am Coll Cardiol. 1993 Oct;22(4 Suppl A):6A-13A. doi: 10.1016/0735-1097(93)90455-a. PMID 8376698
- [Background] He J, Ogden LG, Bazzano LA, Vupputuri S, Loria C, Whelton PK. Risk factors for congestive heart failure in US men and women: NHANES I epidemiologic follow-up study. Arch Intern Med. 2001 Apr 9;161(7):996-1002. doi: 10.1001/archinte.161.7.996. PMID 11295963
- [Background] Kannel WB, Ho K, Thom T. Changing epidemiological features of cardiac failure. Br Heart J. 1994 Aug;72(2 Suppl):S3-9. doi: 10.1136/hrt.72.2_suppl.s3. No abstract available. PMID 7946754
- [Background] Gheorghiade M, Bonow RO. Chronic heart failure in the United States: a manifestation of coronary artery disease. Circulation. 1998 Jan 27;97(3):282-9. doi: 10.1161/01.cir.97.3.282. No abstract available. PMID 9462531
- [Background] Schmidt DE, Shah PK. Accurate detection of elevated left ventricular filling pressure by a simplified bedside application of the Valsalva maneuver. Am J Cardiol. 1993 Feb 15;71(5):462-5. doi: 10.1016/0002-9149(93)90458-o. No abstract available. PMID 8430644
- [Background] Meyer P, Ekundayo OJ, Adamopoulos C, Mujib M, Aban I, White M, Aronow WS, Ahmed A. A propensity-matched study of elevated jugular venous pressure and outcomes in chronic heart failure. Am J Cardiol. 2009 Mar 15;103(6):839-44. doi: 10.1016/j.amjcard.2008.11.045. PMID 19268742
- [Background] Metra M, Ponikowski P, Dickstein K, McMurray JJ, Gavazzi A, Bergh CH, Fraser AG, Jaarsma T, Pitsis A, Mohacsi P, Bohm M, Anker S, Dargie H, Brutsaert D, Komajda M; Heart Failure Association of the European Society of Cardiology. Advanced chronic heart failure: A position statement from the Study Group on Advanced Heart Failure of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2007 Jun-Jul;9(6-7):684-94. doi: 10.1016/j.ejheart.2007.04.003. Epub 2007 May 3. PMID 17481947
- [Background] Killip T 3rd, Kimball JT. Treatment of myocardial infarction in a coronary care unit. A two year experience with 250 patients. Am J Cardiol. 1967 Oct;20(4):457-64. doi: 10.1016/0002-9149(67)90023-9. No abstract available. PMID 6059183